CLINICAL TRIAL: NCT04986761
Title: Patient-reported Outcome Measures (PROMs) Comparing Digital and Conventional Workflows for Treatment With Single-unit Implant Restorations: A Randomized Controlled Trial
Brief Title: PROMs Comparing Digital & Conventional Workflows
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: ITI International Team for Implantology, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MU-DT/PY-IRB 2019/DT146
Record Dates: First submitted 2021-07-01; First posted 2021-08-03 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-08

CONDITIONS: Dental Implant
Keywords: Clinical Research; Dental Implant; Digital Workflow; Patient-Reported Outcome Measures (PROMs); Crowns; Functional Implant Prosthodontic Score (FIPS)

STUDY DESIGN:
Intervention Model Description: Digital and conventional workflows for treatment of implant single crowns, and also the material used.
Who Masked: Outcomes Assessor
Masking Description: Outcomes Assessor received only data without participant group assigned after the intervention was done by a investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Workflows (Experimental): Digital and conventional workflows for treatment of implant single crowns
  Interventions: Procedure: Treatment of implant single crown
- Materials (Experimental): Materials for treatment of implant single crowns (polymer-infiltrated ceramic networks, PICNs and lithium disilicate, LS2).
  Interventions: Procedure: Treatment of implant single crown

INTERVENTIONS:
Procedure: Treatment of implant single crown — Digital or Conventional Workflows for treatment of implant single crown and materials used.

SUMMARY:
This randomized controlled trial (RCT) analyzed monolithic single-unit implant restorations out of lithium disilicate (LS2) or polymer-infiltrated ceramic networks (PICN) in a chairside digital workflow (Test) and a conventional protocol (Control). The primary outcome was subjective patient perception in terms of PROMs comparing digital and conventional impression techniques as well as patients' satisfaction related to the final implant restoration among difference workflows and materials. The secondary outcome was to investigate the objective evaluation by a dental professional applying the functional implant prosthodontic score (FIPS). The null-hypothesis of this RCT was that both workflows and the two materials for the monolithic implant restorations had comparable results with respect to the defined outcomes.

ELIGIBILITY:
Inclusion Criteria:

-The participants are in the age of more than 20 years old and not more than 80 years old.

* The participants who have a transmucosal implant system (Straumann TL RN/WN, Institut Straumann, AG, Basel, Switzerland) placed in single-tooth gap in the area of premolar or molar regions in the maxilla and mandible with existing interproximal and antagonist contacts.
* The participants' general medical health is healthy or has a well-controlled systemic disease.
* The participants' general oral health has shown no sign of infection or unsuccessfully treated diseases such as chronic periodontitis.

Exclusion Criteria:

* The participants who are smoking more than 10 cigarettes per day.
* The participants with pregnancy.
* The participants with a psychiatric disorder
* The participants with a history of radiation therapy at the head and neck area.
* The participants with a history of chemotherapy.
* The participants with bony pathologies such as osseous dysplasia, odontogenic cyst or tumor, etc.

Min Age: 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Patient reported outcome measure (PROM): satisfaction with impression technique via VAS questionnaire | After impression, At first visit within 30 minutes
  After impression-taking, questionnaires were handed out to the participants to evaluate PROMs via visual analog scales (VAS). Six categories were assessed: (1) overall treatment time of impression-taking procedure (0=unsatisfactory to 10=excellent); (2) convenience level of the impression technique (0=unsatisfactory to 10=excellent); (3) anxiety level of impression technique (0=low to 10=high); (4) bad taste and (5) nausea caused by the impression (each 0=no sensation to 10=a lot of sensation); and (6) pain during impression-taking procedure (0=no pain to 10=a lot of pain).
Patient reported outcome measure (PROM): satisfaction with final implant restoration via VAS questionnaire | 1 week after prosthesis delivery
  Patients were requested to score their feeling on screw-retained monolithic implant crowns in a 10cm VAS one week after delivery of the final implant crowns. The level of patients' satisfaction was measured in four categories: (1) perception of the overall treatment outcome (0=unsatisfactory to 10=excellent); (2) opinion on the function of the restoration (0=unsatisfactory to 10=excellent); (3) esthetic perspective (0=unsatisfactory to 10=excellent), and (4) ease of oral hygiene care (0=unsatisfactory to 10=excellent).

SECONDARY OUTCOMES:
Functional implant prosthodontic score (FIPS) | Prosthesis delivery visit, an average of 2 weeks after first visit for impression procedure
  objective evaluation by a dental professional applying the functional implant prosthodontic score (FIPS).

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Mahidol University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Joda T, Bragger U. Patient-centered outcomes comparing digital and conventional implant impression procedures: a randomized crossover trial. Clin Oral Implants Res. 2016 Dec;27(12):e185-e189. doi: 10.1111/clr.12600. Epub 2015 Apr 12. PMID 25864771